CLINICAL TRIAL: NCT06739668
Title: Microtesla Magnetic Therapy (MMT) Treatment of Post-acute Sequelae of SARS CoV-2 (PASC): Controlled Pilot Study
Brief Title: Humanity Neurotech Device Clinical Trial in Adults With Long COVID Cognitive Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Humanity Neurotech Inc. (Unknown)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: STUDY-24-01276
Record Dates: First submitted 2024-12-17; First posted 2024-12-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19 Syndrome; Cognitive Dysfunction
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomization, 2:1, Active to Sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active device (Experimental): The active device will generate a low amplitude magnetic field. 20 participants will be randomized to this arm.
  Interventions: Device: Pascal device
- Sham device (Sham Comparator): The sham device will not generate a low amplitude magnetic field. 10 participants will be randomized to this arm.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Pascal device — The study devices consist of a tabletop Console with user interface and a head-worn applicator (Headset) that is connected via coaxial cable. The Headset is positioned on the head per instructions, and then the study subject powers on the device by pressing the power button and initiates a 15-minute treatment by pressing the start button. LED lights on the console count down during the treatment to indicate time remaining and, once the treatment is complete, the device automatically powers off.
  Arms: Active device
Device: Sham Device — The sham device will look identical to the active device and will have the same indicator lights and sounds, but will not emit magnetic field therapy.
  Arms: Sham device

SUMMARY:
The purpose of this study is to assess the feasibility of an at-home MMT treatment in patients with cognitive dysfunction related to PASC, and to collect data on safety and efficacy to inform the design of larger clinical studies. A prospective randomized controlled study of 30 participants with PASC and moderate to severe cognitive dysfunction. Total study duration will be 8 weeks, including 4 weeks of treatment and 4 weeks of untreated follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English Speaking
* SARS CoV-2 infection as documented by laboratory nucleic acid amplification test or antibody test ≥ 6 months from screening or signed attestation of positive test result
* Experiencing PASC symptoms ≥ 6 months
* Objective cognitive impairment on neuropsychological measures (as defined by a z-score ≥1 standard deviation below the normative mean) in executive functioning
* Individuals of childbearing age agreeing to use a highly effective form of birth control

Exclusion Criteria:

* History of cognitive dysfunction present prior to SARS CoV-2 infection
* Febrile (> 99 F) at the time of the enrollment visit
* Enrollment in another interventional clinical trial in the last 90 days or during the study period
* Recent SARS CoV-2 reinfection in the last 30 days or during the study period
* Recent SARS CoV-2 vaccination in the last 30 days or plans to be vaccinated during the 8 week study period
* Currently taking immunomodulatory medication on an ongoing basis (NSAIDs, corticosteroids, cytokine antagonists, IVIG)
* History of bipolar disorder, psychotic disorder, substance use disorder
* Change in anti-depressant or other psychoactive medication or dose in the last 90 days
* Cranially implanted devices or metal
* Any serious unstable medical or neurologic condition
* History of severe head injury (as defined by loss of consciousness for ≥30 minutes) or stroke in the past 12 months
* Pregnant or plan to become pregnant during the study as indicated by positive pregnancy test
* Serious immune/autoimmune diagnoses prior to SARS-CoV-2 infection
* ME/CFS diagnosis prior to first SARS-CoV-2 infection
* Existing diagnosis of Post-treatment Lyme Disease Syndrome
* Inability to achieve appropriate positioning of the study device on the head

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Successfully Completed Treatments | End of treatment, 4 weeks
  Feasibility of using the device at home will be measured based upon the proportion of successfully completed treatments.

SECONDARY OUTCOMES:
Device comfort | End of treatment, 4 weeks
  Comfort will be assessed using a 5-point Likert scale, full scale from 1-5 with higher scores indicating greater comfort.
Device ease of use | End of treatment, 4 weeks
  Ease of use will be assessed using a 5-point Likert scale, full scale from 1-5 with higher scores indicating greater ease of use.
Clarity of instructions | End of treatment, 4 weeks
  Clarity of instructions will be assessed using a 5-point Likert scale, full scale from 1-5 with high scores indicating greater clarity of instructions.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Cohen Center for Recovery from Complex Chronic Illnesses (CoRE), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.